CLINICAL TRIAL: NCT02109835
Title: Progression of Coronary Atherosclerosis in Asymptomatic Diabetic Subjects: Evaluation of the Role of CT Coronary Angiography and Novel Bio-markers of Endothelial Dysfunction and Vascular Inflammation
Brief Title: Progression of Coronary Atherosclerosis in Asymptomatic Diabetic Subjects
Acronym: PROCEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Cardiac Research Trust (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other); Barnet and Chase Farm Hospitals NHS Trust (Other); Diabetes and Obesity Research Network (Network); Lund University (Other); Health Diagnostic Laboratory, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCRT/3277/PROCEED
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease
Keywords: Diabetes; coronary artery disease; Cardiac computed tomography; Computed tomographics coronary angiography; Plaque progression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum will be separated from the blood sample collected within half an hour. These samples will be labelled with the unique random number assigned to each patient recruited to the study. The link file with the random numbers and patient identifiers will be kept on single computer with restricted access to only members of the research team. Only the completely anonymised samples will be sent to the labs for analysis. 5 mls of whole blood with cells will also be stored.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asymptomatic type 2 diabetes: Patients without previous history of coronary artery disease

SUMMARY:
The purpose of the study is to identify a sub-group of diabetic patients at higher risk of progression of coronary disease and also more likely to suffer from heart attack/angina and heart failure. The total number of patients to be recruited in this study will be 250 with type-2 diabetes but no known heart disease. These patients will have an objective measure of the function of the lining of the arteries, CT scan of the arteries of the heart and an ultrasound scan of the heart and arteries of the neck done at baseline along with blood tests for identification new markers of malfunction of the lining and inflammation of the arteries. Patients will be followed up at 18 months. During the follow-up visit, in addition to the blood tests, the CT scan of the heart arteries and ultrasound of the heart and arteries of the neck will be repeated to assess progression of the non-calcified, calcified and mixed plaques in the coronary arteries.

DETAILED DESCRIPTION:
Hypothesis: We hypothesise that a combination of CT coronary angiography, ultrasound of the heart and of the arteries of the neck, evaluation of expression of genetic markers and bio-markers in the blood will help identify diabetic patients at highest risk of heart disease progression,that can result in angina, heart attacks, heart failure and cardiovascular deaths.

Previous studies using coronary calcium scanning in diabetic patients showed that those with the greatest progression in calcified plaque in the coronary arteries were at the highest risk for heart attacks. However, coronary calcium scans only identify the calcified plaque and are not able to pick up non-calcified, cholesterol rich plaques. Cholesterol rich non-calcified plaques are more often associated witn acute heart attacks. CT coronary angiography can identify both calcified and non-calcified plaques and can therefore add significantly to our predictive ability. Certain chemical substances (biomarkers) measured in blood indicate the severity of plaque burden and inflammation in the coronary arteries. A combination of CT coronary angiography, expression of genetic markers, measure of function of the cells lining the blood vessels and biomarkers can help to identify diabetic patients at highest risk of heart attacks, allowing us to start appropriate risk reduction treatments in those patients. In previous studies with coronary artery calcium, patients suffering from heart attacks were those who also had a higher progression of coronary artery calcium (CAC) score. In diabetics, in particular, patients with poor control of their blood glucose also had greater progression of the CAC score. In order to test the validity of our hypothesis, we have decided to base our study on a population of established diabetics with difficult to control blood pressure, high cholesterol and chronic complications of the small blood vessels, i.e. involvement of the retina (back of the eye) and peripheral nerves as well as protein in the urine. Patients with chronic complications of diabetes are known to have higher incidence of heart disease as well.

Methodology and Timetable: Patients will be recruited from Diabetes clinics of NHS hospitals in North West London.

If eligible for the trial, an informed consent will be obtained from the patients and their general practitioner will be subsequently informed about their participation in the trial. Once recruited into the trial, a CT coronary angiogram (CTCA, CT of the arteries of the heart), ultrasound scan of the heart and carotid arteries of the neck as well as a measure of endothelial function will be performed at the Wellington Hospital in St. Johns Wood, London within 1-2 weeks. At the same time, blood samples will also be obtained for bio-markers. A report of the CTCA will then be forwarded to the consultant in-charge of the patient's care as well as to the GP.

If a narrowing of moderate degree (70%) is noted on the CT angiogram, the patient will then be brought back to the Wellington Hospital within 2 weeks for a heart perfusion scan which evaluates the relative discrepancies in flow of blood to the heart muscle and helps plan further management.

If there is significant reduction in blood flow noted in the perfusion scan,patients will be referred back to the consultants for further clinical management.

During their first visit to the Wellington Hospital for the CT scan, blood samples will be taken and stored on-site for biomarker analysis.

Patients will be followed up after 18 months from the time of recruitment into the trial,when a second CTCA, ultrasound of the arteries of the neck will be performed to assess the degree of progression of calcium and cholesterol deposits within the coronary arteries and thickness of the lining of the arteries in the neck in addition to blood sample collection for bio-markers.

Patients with significant narrowing of coronary arteries (>70%) requiring a stent to be inserted in the first scan will be excluded from follow up. Patients with normal coronary arteries on the initial scan also will be excluded from the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Established T2DM with or without micro-vascular complications of diabetes (retinopathy, peripheral neuropathy and/or micro-albuminuria)

No history of coronary artery disease (CAD)

Exclusion Criteria:

* 1. Estimated GFR <45 2. Pregnant women 3. Age < 35 years 4. Atrial fibrillation 5. Known allergy to iodine contrast 6. CAC score >1000 Agatston Units

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes recruited from hospital clinics and one community faith based cardiovascular disease prevention clinic run under the aegis of a lipidologist
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Greater than 20% increase in plaque volume | 18 months
  Plaque volume will be measured by both manual and semi-quantitative methods

SECONDARY OUTCOMES:
Greater than 20% increase in coronary artery calcium score | 18 months
  Coronary artery calcium scoring will be performed using a semi-quantitative method.

OTHER OUTCOMES:
Correlation between increase in plaque volume with levels of biomarkers | 18 months
  Correlate plaque progression with various bio-markers
Correlation between carotid IMT measurements and coronary plaque | 18 months
  Once at baseline and then during follow-up
Incidence of major adverse cardiovascular events (MACE) during the 18-month follow-up period. MACE is defined as incidence of cardiac death, non-fatal myocardial infarction, STEMI and NSTEMI, unstable angina, late revascularization and onset of angina | 18 months
  Through questionnaires and medical records

CONTACTS AND LOCATIONS:
Overall Officials: Roby Rakhit, MD FRCP, Study Chair — Royal Free Hospital NHS Foundation Trust; Avijit Lahiri, MRCP FACC, Study Director — Wellington Hospital; Daniel Darko, MRCP, Principal Investigator — Central Middlesex Hospital; Mark Cohen, PhD FRCP, Principal Investigator — Barnet Hospital; Rajiv A Amersey, MD FRCP, Principal Investigator — Whipps Cross Hospital; Sarita Naik, DM MRCP, Principal Investigator — University College London Hospital
Locations (5):
- United Kingdom (5):
  - Central Middlesex Hospital, London, Middlesex
  - Barts Health NHS Trust, London
  - Barnet Hospital, London
  - University College London Hospitals, London
  - Royal Free Hospital, London

REFERENCES:
- [Background] Anand DV, Lim E, Lahiri A, Bax JJ. The role of non-invasive imaging in the risk stratification of asymptomatic diabetic subjects. Eur Heart J. 2006 Apr;27(8):905-12. doi: 10.1093/eurheartj/ehi441. Epub 2005 Aug 8. PMID 16087647
- [Background] Anand DV, Lahiri A, Lim E, Hopkins D, Corder R. The relationship between plasma osteoprotegerin levels and coronary artery calcification in uncomplicated type 2 diabetic subjects. J Am Coll Cardiol. 2006 May 2;47(9):1850-7. doi: 10.1016/j.jacc.2005.12.054. Epub 2006 Apr 19. PMID 16682312
- [Background] Anand DV, Lim E, Darko D, Bassett P, Hopkins D, Lipkin D, Corder R, Lahiri A. Determinants of progression of coronary artery calcification in type 2 diabetes role of glycemic control and inflammatory/vascular calcification markers. J Am Coll Cardiol. 2007 Dec 4;50(23):2218-25. doi: 10.1016/j.jacc.2007.08.032. Epub 2007 Nov 19. PMID 18061069
- [Background] Fredrikson GN, Anand DV, Hopkins D, Corder R, Alm R, Bengtsson E, Shah PK, Lahiri A, Nilsson J. Associations between autoantibodies against apolipoprotein B-100 peptides and vascular complications in patients with type 2 diabetes. Diabetologia. 2009 Jul;52(7):1426-33. doi: 10.1007/s00125-009-1377-9. Epub 2009 May 12. PMID 19448981
- [Background] Jeevarethinam A, Venuraju S, Weymouth M, Atwal S, Lahiri A. Carotid intimal thickness and plaque predict prevalence and severity of coronary atherosclerosis: a pilot study. Angiology. 2015 Jan;66(1):65-9. doi: 10.1177/0003319714522849. Epub 2014 Feb 26. PMID 24576983
- [Derived] Venuraju SM, Lahiri A, Jeevarethinam A, Cohen M, Darko D, Nair D, Rosenthal M, Rakhit RD. Duration of type 2 diabetes mellitus and systolic blood pressure as determinants of severity of coronary stenosis and adverse events in an asymptomatic diabetic population: PROCEED study. Cardiovasc Diabetol. 2019 Apr 23;18(1):51. doi: 10.1186/s12933-019-0855-8. PMID 31014330